CLINICAL TRIAL: NCT06135545
Title: Comparing the Postoperative Analgesic Effects of Bupivacaine Liposome Serrate Anterior Plane Block (SAPB) Versus Traditional Thoracic Paravertebral Block (TPVB): A Randomized, Double-blinded Non-inferiority Clinical Trial
Brief Title: Bupivacaine Liposome Serrate Anterior Plane Block vs Traditional Thoracic Paravertebral Block
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Shiyou Wei (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023LY0519
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
Keywords: Serratus anterior plane block; Thoracic paravertebral block; Liposomal bupivacaine; Video-assisted thoracoscopic surgery; Postoperative pain
MeSH Terms: conditions — Lung Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded non-inferiority clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T Group (Experimental): The T group used liposomal bupivacaine for ultrasound-guided serratus anterior plane block.
  Interventions: Combination Product: Bupivacaine Liposome SAPB
- C Group (Active Comparator): The C group used traditional ropivacaine for ultrasound-guided paravertebral nerve block.
  Interventions: Combination Product: Traditional TPVB

INTERVENTIONS:
Combination Product: Bupivacaine Liposome SAPB — Dilute 266mg of bupivacaine liposome with saline solution to 30ml.The patients are placed in the lateral position and the probe is placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The investigators count the ribs inferiorly and laterally, until The investigators identify the fifth rib in the midaxillary line. The latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscles (deep and inferior) are then easily identifiable by ultrasound overlying the fifth rib.
  Other Names: Bupivacaine Liposome Serrate Anterior Plane Block(SAPB)
  Arms: T Group
Combination Product: Traditional TPVB — The TPVB was recommended by the American Society of Anesthesiologists.The transducer is placed sagitally over a transverse process(TP), placing it at the center of the ultrasound image. Alternatively, the space in-between two adjacent transverse processes may be positioned at the center. The needle is inserted using an out-of-plane technique and advanced until the central TP is contacted, or else the cranial of the two, with no or minimal angulation in the sagittal plane or the transversal plane. Subsequently, the needle is walked off the TP into the TPV space and advanced 1 to 1.5 cm beyond the TP without further visualizing the needle tip on ultrasound. Entering of the needle tip into the TPV space can result in a loss of resistance to normal saline and by visualizing anterior displacement of the pleura upon injection. Select the fifth TP as the insertion point, and inject 20ml of 0.5% ropivacaine (Hengrui, Jiangsu) into the TPV space.
  Other Names: Traditional Thoracic Paravertebral Block(TPVB)
  Arms: C Group

SUMMARY:
In this study, patients will receive bupivacaine liposome serratus anterior plane block or ropivacaine paraspinal block to manage postoperative pain. Follow-up visits will be conducted to investigate the patient's postoperative pain and recovery quality. The investigators hypothesize that the simple and safe serratus anterior plane block with a novel long-acting local anesthetic (bupivacaine liposome) has analgesic efficacy and recovery quality that is not inferior to the currently commonly used bupivacaine paraspinal block.

DETAILED DESCRIPTION:
Extensive research suggests that paravertebral block can replace thoracic epidural anesthesia as the "gold standard" for thoracic surgery pain relief. However, this technique is more challenging than the fascial plane block and carries the risk of damaging the pleura or spinal nerve roots. The serratus anterior plane block (SAPB) was refined by Blanco et al. in 2013 and is a new, safe regional anesthesia technique that can block the lateral cutaneous branches of the intercostal nerves from T2 to T9, as well as the long thoracic nerve, providing intraoperative and postoperative pain relief for surgeries in this area. A meta-analysis has reported that it can be an alternative regional anesthesia method to paravertebral and intercostal nerve blocks, and is technically safer, more effective, easier to perform, and may have fewer adverse reactions, making it more favored by clinicians. However, a recent network meta-analysis of regional block techniques in thoracic surgery suggested that, in terms of postoperative pain scores at 24 hours, SAPB can relieve pain but is slightly inferior to paravertebral block.

The duration of action of currently used local anesthetics is short. Although various adjuvants have been proposed, such as dexamethasone and dexmedetomidine, there are currently no drugs approved by the FDA that reliably extend the duration of local anesthetics beyond 24 hours (PMID: 27749354). Liposomal encapsulation of bupivacaine can extend the release time of local anesthetics to 72-96 hours (PMID: 23229686, 28120158), with the potential to reduce pain scores at 72 hours postoperatively (PMID: 22067185). Liposomal bupivacaine (Hengrui, Jiangsu) is also the first long-acting local anesthetic currently on the market in China, sparking new hope for anesthesiologists to better manage postoperative pain.

This study hypothesizes, from a clinical perspective, that the use of long-acting local anesthetic liposomal bupivacaine in a simplified and safe serratus anterior plane block technique for regional pain relief postoperatively is not inferior to the widely accepted gold standard for thoracic pain relief-paravertebral block with ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral thoracoscopic lung surgery.
* Age between 18 and 75 years old.
* American Society of Anesthesiologists (ASA) classification I to III.

Exclusion Criteria:

* Contraindications to nerve block: puncture site infection, local anesthetic allergy, coagulation disorders or risk of bleeding.
* Hepatic or renal dysfunction.
* Pregnant, breastfeeding, possibility of pregnancy or planned pregnancy.
* Use of analgesic drugs before surgery or history of chronic pain or opioid abuse.
* Patients who refuse to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-10-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative NRS pain score at 24 hours | 24 hours after the surgery
  Postoperative numeric rating scales pain score at 24 hours after the surgery. Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.

SECONDARY OUTCOMES:
Postoperative QoR-15 | 24 to 72 hours after the surgery
  The 15-item quality of recovery(QoR-15) after the surgery. The QoR-15 scale is a global measurement of postoperative recovery, consisting of 15 items with 10 points each, with a total score ranging from 0 (QoR very poor) to 150 (QoR very good).
Cumulative opioid consumption after surgery | 72 hours after the surgery
  Cumulative opioid consumption after surgery
AUC of postoperative pain score | 72 hours after the surgery
  Area under the curve(AUC) of pain score 72 hours after surgery
Postoperative NRS pain score | 1h, 6h, 48h, 72h after the surgery, separately.
  Pain scores at other time points except for the primary outcome. Postoperative pain severity at rest and movement measured using a numerical rating scale(NRS) at 24 h. The numerical rating scale (NRS) is a line with numbers from 0 to 10 are spaced evenly across the page. And the NRS is bounded at the left-most end with "no pain" and at the right-most end with "worst pain imaginable". Pain levels below "4" are considered mild, "4-7" is moderate pain, and anything above "7" is considered severe pain. Patients are instructed to circle the number that represents the amount of pain that they are experiencing at the time of the evaluation. The movement status refers to maximum mobility of the upper arm of the surgical side. Remedial pain relief measures are initiated when the Numeric Rating Scale (NRS) score exceeds 4.

OTHER OUTCOMES:
The number of patients receiving rescue analgesia. | 24 to 72 hours after the surgery
  The number of patients receiving rescue analgesia.
Number of patients with nausea and vomiting | 24 to 72 hours after the surgery
  Number of patients who experienced nausea and vomiting after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Song, MD., Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Chong M, Berbenetz N, Kumar K, Lin C. The serratus plane block for postoperative analgesia in breast and thoracic surgery: a systematic review and meta-analysis. Reg Anesth Pain Med. 2019 Oct 23:rapm-2019-100982. doi: 10.1136/rapm-2019-100982. Online ahead of print. PMID 31649029
- [Background] Sandeep B, Huang X, Li Y, Xiong D, Zhu B, Xiao Z. A comparison of regional anesthesia techniques in patients undergoing video-assisted thoracic surgery: A network meta-analysis. Int J Surg. 2022 Sep;105:106840. doi: 10.1016/j.ijsu.2022.106840. Epub 2022 Aug 24. PMID 36030040
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] Hu D, Onel E, Singla N, Kramer WG, Hadzic A. Pharmacokinetic profile of liposome bupivacaine injection following a single administration at the surgical site. Clin Drug Investig. 2013 Feb;33(2):109-15. doi: 10.1007/s40261-012-0043-z. PMID 23229686
- [Background] Rice D, Heil JW, Biernat L. Pharmacokinetic Profile and Tolerability of Liposomal Bupivacaine Following a Repeated Dose via Local Subcutaneous Infiltration in Healthy Volunteers. Clin Drug Investig. 2017 Mar;37(3):249-257. doi: 10.1007/s40261-017-0495-2. PMID 28120158
- [Background] Krediet AC, Moayeri N, van Geffen GJ, Bruhn J, Renes S, Bigeleisen PE, Groen GJ. Different Approaches to Ultrasound-guided Thoracic Paravertebral Block: An Illustrated Review. Anesthesiology. 2015 Aug;123(2):459-74. doi: 10.1097/ALN.0000000000000747. PMID 26083767
- [Result] Ding W, Chen Y, Li D, Wang L, Liu H, Wang H, Zeng X. Investigation of single-dose thoracic paravertebral analgesia for postoperative pain control after thoracoscopic lobectomy - A randomized controlled trial. Int J Surg. 2018 Sep;57:8-14. doi: 10.1016/j.ijsu.2018.07.006. Epub 2018 Jul 26. PMID 30056127